CLINICAL TRIAL: NCT04712578
Title: Influence of Caffeinated and Non-caffeinated Pre-workout Supplements on Resistance Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Legion Athletics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB2020-813; 20-1299 (Other: Texas Tech University Sponsored Projects)
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Resistance Training; Caffeine; Dietary Supplements
Keywords: caffeine; resistance training; resistance exercise; pre-workout supplement; dietary supplements

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled crossover trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All investigators will be blinded to the caffeinated vs. non-caffeinated supplement (i.e., these were provided by the manufacturer in a blinded manner). Select study investigators who will not be involved in assessing outcomes will formulate the placebo supplement and be responsible for dispensing all supplements to participants. Supplements will be provided to participants in opaque containers to maintain blinding. All investigators involved in assessing outcomes will also remain blinded and will not be involved in handling or dispensing the supplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeinated Pre-workout Supplement (Experimental): This arm will consist of ingestion of the commercially available, caffeinated Pulse pre-workout, manufactured by Legion Athletics, Inc.
  Interventions: Dietary Supplement: Caffeinated pre-workout supplement
- Non-Caffeinated Pre-Workout Supplement (Active Comparator): This arm will consist of ingestion of the commercially available, non-caffeinated Pulse pre-workout, manufactured by Legion Athletics, Inc.
  Interventions: Dietary Supplement: Non-caffeinated pre-workout supplement
- Placebo (Placebo Comparator): This arm will consist of a flavor-matched placebo beverage without the active components contained in the supplements administered in the other study arms.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeinated pre-workout supplement — The intervention will consist of consuming a standardized meal followed by one serving of the commercially available Pulse caffeinated pre-workout supplement (Legion Athletics, Inc.).
  Other Names: Legion Athletics Pulse Pre-workout Supplement
  Arms: Caffeinated Pre-workout Supplement
Dietary Supplement: Non-caffeinated pre-workout supplement — The intervention will consist of consuming a standardized meal followed by one serving of the commercially available Pulse non-caffeinated pre-workout supplement (Legion Athletics, Inc.).
  Other Names: Legion Athletics Pulse Pre-workout Supplement
  Arms: Non-Caffeinated Pre-Workout Supplement
Dietary Supplement: Placebo — The intervention will consist of consuming a standardized meal followed by a placebo beverage.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled crossover trial examining the effects of caffeinated and non-caffeinated pre-workout supplements on resistance exercise performance. Resistance-trained adults will be randomly assigned to complete three study conditions (caffeinated pre-workout, non-caffeinated pre-workout, and placebo) in one of the six possible condition orders. During each condition, participants will report to the laboratory for ingestion of the assigned beverage and subsequent muscular performance testing. Major performance outcomes will be force production variables from a mechanized squat device and maximal strength and muscular endurance on the bench press and leg press exercises.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40;
* Body mass between 50 - 100 kg (110-220 lb)
* Generally healthy (defined as an absence of any disease or medical condition which could potentially be negatively affected by consumption of the commercially available dietary supplements or performance of exercise, including but not limited to musculoskeletal or cardiovascular diseases).
* Resistance-trained, defined as completing 2+ resistance training sessions per week for at least three months prior to screening.
* Participants must have reported regular training of the lower body through a multi-joint exercise such as the squat or leg press at least once weekly during the three-month period prior to screening.
* Participants must have reported regular training of the bench press or chest press variation at least once weekly during the three-month period prior to screening.
* Female participants will be required to bench press ≥ 0.5 x body mass and leg press ≥ 1.75 x body mass during initial 1RM assessments to be eligible for this study.
* Male participants will be required to bench press ≥ 1.0 x body mass and leg press ≥ 3.0 x body mass to be eligible.
* Regular caffeine consumption (due to the presence of caffeine in the commercially available dietary supplement). This will be defined as an average self-reported daily intake of 250+ mg of caffeine, which is equivalent to approximately 2.5 cups of coffee.

Exclusion Criteria:

* Failing to meet any of the aforementioned inclusion criteria.
* Pregnant or breastfeeding (for female participants)
* Taking prescription medication which could reasonably make participation unsafe for the participant or influence study outcomes
* An inability to complete resistance exercise due to injury or medical condition
* Self-reported caffeine sensitivity, as indicated by unwanted side effects when caffeine is consumed.
* Allergy to any of the ingredients in the test beverages or standardized breakfast.
* Current use of anabolic steroids
* Presence of a pacemaker or other implanted electrical device.
* Unwillingness to wear the provided surgical mask during all testing procedures.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Isometric Peak Force Production | Approximately 35 minutes after beverage ingestion in each condition.
  Peak isometric force produced on a mechanical squat device at an 120-degree knee angle.
Isometric Rate of Force Development | Approximately 35 minutes after beverage ingestion in each condition.
  Rate of force development produced on a mechanical squat device at an 120-degree knee angle.
Isokinetic Peak Concentric Force Production | Approximately 40 minutes after beverage ingestion in each condition.
  Peak concentric force produced during isokinetic testing on a mechanical squat device.
Isokinetic Peak Eccentric Force Production | Approximately 40 minutes after beverage ingestion in each condition.
  Peak eccentric force produced during isokinetic testing on a mechanical squat device.
Maximal Strength on Bench Press Exercise | Approximately 65 minutes after beverage ingestion in each condition.
  One-repetition maximum for the barbell bench press exercise.
Muscular Endurance on Bench Press Exercise | Approximately 70 minutes after beverage ingestion in each condition.
  Repetitions to failure on the bench press exercise, using a load corresponding to 0.4 times body mass for females and 0.75 times body mass for males.
Maximal Strength on Leg Press Exercise | Approximately 95 minutes after beverage ingestion in each condition.
  One-repetition maximum for the plate-loaded leg press exercise.
Muscular Endurance on Leg Press Exercise | Approximately 100 minutes after beverage ingestion in each condition.
  Repetitions to failure on the leg press exercise, using a load corresponding to 1.5 times body mass for females and 2.5 times body mass for males.

SECONDARY OUTCOMES:
Subjective Ratings of Energy | Five total assessments in each condition. Immediately prior to: beverage ingestion, isometric exercise testing, bench press testing, and leg press testing. Also, immediately after leg press testing.
  Subjective rating of energy as indicated by visual analog scale (0 to 100, with a higher value indicating a higher rating of energy).
Subjective Ratings of Focus | Five total assessments in each condition. Immediately prior to: beverage ingestion, isometric exercise testing, bench press testing, and leg press testing. Also, immediately after leg press testing.
  Subjective rating of focus as indicated by visual analog scale (0 to 100, with a higher value indicating a higher rating of focus).
Subjective Ratings of Fatigue | Five total assessments in each condition. Immediately prior to: beverage ingestion, isometric exercise testing, bench press testing, and leg press testing. Also, immediately after leg press testing.
  Subjective rating of fatigue as indicated by visual analog scale (0 to 100, with a higher value indicating a higher rating of fatigue).

OTHER OUTCOMES:
Participant Identification of Beverage | At the very end of each condition (i.e., approximately 105 minutes after beverage ingestion in each condition; exact time of assessment may vary based on duration of exercise performance testing for each participant).
  At the end of each exercise session (i.e., after leg press testing has concluded), participants will be asked to identify the test beverage they believe they received.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States